CLINICAL TRIAL: NCT03480490
Title: Evaluation and Outcome of Para-pneumonic Effusion Among Children Attending Assuit University Pediatric Hospital
Brief Title: Evaluation and Outcome of Para-pneumonic Effusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Rashad Ahmed Hassan, Principle investigator, Assiut University
Other Study IDs: EOPE
Record Dates: First submitted 2018-03-19; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pleural fluid C-reactive protein — C-reactive protein is an acute phase protein that is synthesized by the liver in response to various stimuli.
  The pleural fluid c-reactive protein levels are likely to reflect the serum levels because the presence of c-reactive protein in the pleural fluid may be due to increased diffusion from the blood as a result of inflamed capillary leakage.
  Pleural c-reactive protein has been proposed as a specific biomarker for the differential diagnosis of pleural effusions and reportedly exhibits higher sensitivity and specificity than serum c-reactive protein.
  c-reactive protein can be considered a good candidate due to its 1000-fold elevation in response to infection and the positive correlation between the serum and pleural c-reactive protein levels.
  Pleural fluid c-reactive protein level was significantly higher in exudates than that in transudative effusion.

SUMMARY:
Pleural effusion is the accumulation of excess fluid in the pleural cavity, which results in disturbance of the equilibrium between vascular hydrostatic and oncotic pressures. The underlying causes of pleural effusion include pleural inflammation or infection, congestive heart failure, lymphatic drainage blockage and malignancy.A parapneumonic effusion is a pleural effusion associated with lung infection. Early in the course of parapneumonic effusion, the pleura becomes inflamed with leakage of cellular elements, protein, and fluid into the pleural space, forming the effusion. Subsequent bacterial invasion results in a frank empyema, the presence of which often requires thoracentesis.

DETAILED DESCRIPTION:
A delay in the diagnosis and initiation of proper therapy for infectious effusions leads to increases in the complication rate. These delays are more common in patients with coexisting heart failure or malignancy.In fact, pleural effusion manifestations are alerting signs of pain, dyspnea, and the signs of respiratory failure due to compression of the lungs.

Other signs include tachypnea, decreased percussion, and decreased respiratory sounds. The most common cause of pleural effusion in children is parapneumonic effusion or purulent empyema.

Although the prevalence of pleural effusion is high in children, its mortality rate is low . According to the studies performed in the United States, parapneumonic effusion is known as the most common underlying cause of pleural effusion in 50% to 70% of the cases . Congenital heart diseases include 5-15% of the causes and malignancies are the rare reasons of effusion.

In general, effusions may be transudate or exudate and examination of the pleural fluid is necessary to differentiate them. Exudate is confirmed by the presence of at least one of the following criteria; pleural effusion concentration higher than half of the serum protein level, pleural effusion protein level more than 3 g/dL, pleural effusion lactate dehydrogenase higher than 200 U, pH lower than 7.2, and glucose lower than 40.

C-reactive protein is an acute phase protein that is synthesized by the liver in response to various stimuli.The induction of C-reactive protein synthesis in the liver is triggered by the production of Interleukin-6 and Tumor Necrosis Factor-alpha by local pleural cells.

The pleural fluid C-reactive protein levels are likely to reflect the serum levels because the presence of C-reactive protein in the pleural fluid may be due to increased diffusion from the blood as a result of inflamed capillary leakage.

Pleural C-reactive protein has been proposed as a specific biomarker for the differential diagnosis of pleural effusions and reportedly exhibits higher sensitivity and specificity than serum C-reacive protein. C-reactive protein can be considered a good candidate due to its 1000-fold elevation in response to infection and the positive correlation between the serum and pleural C-reactive protein levels. Pleural fluid C-reactive protein level was significantly higher in exudates than that in transudative effusion.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted upon patients(male and females),from 1 month to 18 years with para-pneumonic effusion at assuit university pediatric hospital from January to june 2019 after taking consents.

Exclusion Criteria:

* age: >18 years old congenital heart disease lymphatic drainage blockage post traumatic pleural effusion renal diseases hepatic diseases neoplastic diseases

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study was conducted on patients with para-pneumonic effusion who were admitted to the Assiut University Pediatrics Hospital in the period between january 2019 and january 2020.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
cure rate from effusion | baseline
  to evaluate the cure rate from para-pneumonic effusion among children

CONTACTS AND LOCATIONS:
Overall Officials: Yasser F Abdel-raheim, PhD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Adeoye PO, Johnson WR, Desalu OO, Ofoegbu CP, Fawibe AE, Salami AK, Fadeyi A, Akin-Dosumu AA, Rasheedat IM; Ilorin Pleural Effusion Study Group. Etiology, clinical characteristics, and management of pleural effusion in Ilorin, Nigeria. Niger Med J. 2017 Mar-Apr;58(2):76-80. doi: 10.4103/0300-1652.219349. PMID 29269986